CLINICAL TRIAL: NCT02353546
Title: Managing Cancer and Living Meaningfully (CALM): Phase 2b Pilot Randomized Psychotherapy Trial in Patients With Advanced Cancer
Brief Title: CALM Phase 2b Pilot
Acronym: CALM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHN 09-0855-C; MOP 106473 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Depression
Keywords: affective symptoms; cancer; depression; palliative care; pilot trial; psychotherapy
MeSH Terms: conditions — Depression; Affective Symptoms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CALM (Experimental): Patients assigned to the intervention arm will receive 3-6 CALM therapy sessions over 3-6 months delivered by a trained therapist at our center.
  Interventions: Behavioral: CALM
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: CALM
  Arms: CALM

SUMMARY:
Managing Cancer And Living Meaningfully (CALM) is a brief psychotherapy designed to alleviate distress in advanced cancer. In an earlier intervention-only pilot trial, CALM was associated with reductions in depressive symptoms and death anxiety and an increase in spiritual wellbeing. The purpose of this study is to assess the feasibility of a large-scale randomized controlled trial (RCT) of CALM and to identify preliminary effects in advanced cancer. This phase 2b pilot RCT employed intervention and usual care arms with 3 and 6 month follow-ups. The primary outcome was depressive symptoms (PHQ-9) and secondary outcomes included diagnosis of major depression (SCID), death anxiety, attachment security and spiritual wellbeing. Multilevel regression was used to compare change over time between groups. 60 patients with advanced cancer will be recruited from the Princess Margaret Cancer Centre, Toronto, Canada, and equally randomized into intervention and usual care conditions.

DETAILED DESCRIPTION:
Abstract

Background Managing Cancer And Living Meaningfully (CALM) is a brief individual psychotherapy for patients with advanced cancer. In an intervention-only phase 2a trial, CALM showed promising results, leading to the present 2b pilot, which introduces procedures for randomisation and improved rigour in preparation for a phase 3 randomised controlled trial (RCT).

Aims To test trial methodology and assess feasibility of a confirmatory RCT.

Design A parallel-arm RCT (intervention vs usual care) with 3 and 6-month follow-ups. Assessment of feasibility included rates of consent, randomisation, attrition, intervention non-compliance and usual care contamination. Primary outcome: depressive symptoms (Patient Health Questionnaire-9; PHQ-9). Secondary outcomes: major depressive disorder (MDD), generalised anxiety, death anxiety, spiritual well-being, attachment anxiety and avoidance, self-esteem, experiential avoidance, quality of life and post-traumatic growth. Bayesian conjugate analysis was used in this low-powered setting.

Setting/participants 60 adult patients with advanced cancer from the Princess Margaret Cancer Centre.

Trial registration number NCT02353546.

http://dx.doi.org/10.1136/bmjspcare-2015-000866

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Fluent in English
* Confirmed diagnosis of Stage IIIB or IV lung cancer, Stage III or IV ovarian cancer, Stage IV endocrine, breast, gastrointestinal, genitourinary or gynecologic cancer, or pancreatic cancer at any stage

Exclusion Criteria:

* Short Orientation-Memory-Concentration Test (score of <20)
* Individuals receiving in-hospital psychiatric or psychological treatment at the time of recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | 6-months

SECONDARY OUTCOMES:
Major Depression Structured Clinical Interview for DSM Disorders (SCID) | 6-months
  DSM: Diagnostic and Statistical Manual of Mental Disorders (APA, 2000)
Generalized Anxiety Disorder-7 (GAD-7) | 6-months
Death and Dying Distress Scale (DADDS) | 6-months
Functional Assessment of Chronic Illness Therapy-Spiritual Well-being Scale (FACIT-Sp-12) | 6-months
Modified Experiences in Close Relationships (ECR M-16) | 6-months
Rosenberg Self-esteem Scale (RSES) | 6-months
Acceptance and Action Questionnaire-II (AAQ-II) | 6-months
Quality of Life at the End of Life-Cancer Scale (QUAL-EC) | 6-months
Posttraumatic Growth Inventory (PTGI) | 6-months

CONTACTS AND LOCATIONS:
Overall Officials: Gary Rodin, Principal Investigator — University Health Network, Toronto; Sarah Hales, Principal Investigator — University Health Network, Toronto; Chris Lo, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Result] Lo C, Hales S, Chiu A, Panday T, Malfitano C, Jung J, Rydall A, Li M, Nissim R, Zimmermann C, Rodin G. Managing Cancer And Living Meaningfully (CALM): randomised feasibility trial in patients with advanced cancer. BMJ Support Palliat Care. 2019 Jun;9(2):209-218. doi: 10.1136/bmjspcare-2015-000866. Epub 2016 Jan 19. PMID 26787360
- See also: Publication in BMJ Supportive and Palliative Care — https://spcare.bmj.com/content/bmjspcare/9/2/209.full.pdf